CLINICAL TRIAL: NCT02551289
Title: MRI Assessment in Newly Diagnosed Coeliac Disease and Following Gluten-free Diet Treatment
Brief Title: MAgnetic Resonance Imaging in COeliac Disease
Acronym: MARCO
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); University of Salerno (Other)
Responsible Party: Sponsor
Other Study IDs: 14MP002
Record Dates: First submitted 2015-09-08; First posted 2015-09-16 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Celiac Disease; Coeliac Disease; Celiac Sprue; Gluten Enteropathy
Keywords: MRI; Gluten; Imaging; Enteropathy-Associated T-Cell Lymphoma
MeSH Terms: conditions — Celiac Disease; Enteropathy-Associated T-Cell Lymphoma | interventions — Diet, Gluten-Free

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients newly diagnosed with Coeliac disease before starting treatment with a gluten free diet
  Interventions: Other: Gluten free diet
- Healthy volunteers: Participants who do not meet criteria for a clinical diagnosis of Coeliac disease as determined by screening blood sample.

INTERVENTIONS:
Other: Gluten free diet — Patients will follow a gluten free diet
  Groups: Patients

SUMMARY:
One in 100 people suffers from coeliac disease. It affects the lining of the bowel and causes many symptoms such as diarrhoea, wind, stomach pain, constipation and nausea. The only treatment so far is a strict glutenfree diet for life which reverses the bowel damage and often improves symptoms. Up to 25% of patients however may have persistent symptoms despite the gluten free diet but the reasons for this are not clear.

This research aims to help us understand how the gluten free diet works. Investigators will use medical imaging (magnetic resonance imaging or MRI) to measure the volumes of fluid in the small bowel, the size of the large bowel and the time it takes for foods to go through the entire bowel in patients who have just been diagnosed with coeliac disease by their hospital doctor. Investigators will also carry out a breath test and collect a stool sample for basic analysis of the stool bacteria.

Investigators will also collect questionnaires about their feelings and their bowel habits and will try to see how the MRI measurements relate to the patients' symptoms. Investigators will observe how all these measures change after one year of the gluten free diet that doctors will have prescribed as part of the coeliac patients' standard care. As such there is no dietary intervention in this study, investigators will simply study changes in the patients due to their standard treatment. Investigators will also look at a matched group of healthy volunteers to gather a likely reference range of the measurements. This research will be carried out in Nottingham with the help of the specialist coeliac clinics and it will last 3 years. There is a dedicated Coeliac Patient Public Involvement group who have helped plan this study.

DETAILED DESCRIPTION:
Hypotheses of the study

Based on the investigators' pilot data and on the literature available, this study aims to test the main hypotheses that in adults newly diagnosed with coeliac disease treatment with GFD will:

1. reduce the water content of the fasting small bowel
2. reduce the volume of the fasting colon
3. increase whole gut transit time

Objectives of the study

The specific objectives of the study are therefore to quantify any change following treatment with a gluten-free diet (GFD) in:

1. the water content of the fasting small bowel
2. fasting colon volume
3. whole gut transit time in adults newly diagnosed with coeliac disease using non-invasive MRI Co-variates of interest

During this study investigators will measure a series of exploratory co-variates of interest at diagnosis and at 12 months follow-up:

1. BMI
2. Gastrointestinal symptoms (Bristol Stool diary for a week, HAD, PHQ-15, IBSS, QOL, GI symptoms VAS scales )
3. Marsh grading of D2 segment duodenal biopsies (defined as routine clinical assessment in NUH)
4. Fasting breath hydrogen
5. Serology values (tTG, EMA)
6. Faecal microbiota and short chain fatty acids

In a subgroup analysis, investigators will describe associations (if any) between the MRI outcomes and these co-variates:

1. before treatment,
2. after treatment and
3. differences between the two.

The latter will represent the most useful analysis. By using the after treatment measure as the outcome and the before treatment measure as a covariate this will be mathematically equivalent to analysing the change with treatment (adjusted for baseline).

Parallel Healthy Volunteers group This study will also include a parallel pilot study healthy volunteers (HVs) frequency matched for age (in 20 years bands) and gender to provide descriptive statistics on a likely reference range for the healthy population to inform the design of future studies.

A pilot study in 36 newly diagnosed coeliac disease patients before and after a gluten-free diet.

University based

Pilot study on patients:

There is no data available to estimate the size of the change in water content of the fasting small bowel in patients hence this is a pilot study.

The investigators' own MRI pilot data in n=20 untreated, newly diagnosed coeliac patients showed a fasting small bowel water content of (mean ± SD) 202 ± 115 ml volume. We can predict that we should be able to detect a change of 40% (or a reduction of 80 ml volume) after gluten free diet with a power of 90% and a Type I error probability of 0.05 using n=24 patients in a paired study design. This is considered a clinically significant change after gluten free diet; this change reflects twice the level of normal control values of 65 ± 43 ml volume. Investigators plan to recruit n=36 to allow for dropouts and to increase power also for secondary outcomes.)

Pilot study on healthy volunteers (HVs):

For exploratory purposes and to provide pilot reference data for the design of future studies, investigators aim to collect data on 36 HVs 36 patients and 36 healthy volunteers.

Pilot study in coeliac disease:

Investigations include:

1. Magnetic Resonance Imaging - 2 scans 12 months apart
2. Self-administered symptom questionnaires
3. Stool sample
4. Hydrogen breath test The patients will have had a biopsy and serology as part of their standard care. The healthy volunteers will undergo only the blood sample as part of screening with no biopsy taken.

Duration of study = 36 months. Duration of study for each participant = around 12 months. Follow-up of participants will stop after 12 months if they fail to receive the subsequent MRI scan There is no randomisation or blinding as this is a simple pilot study. Primary endpoint

1. Fasting small bowel water content (SBWC) measured in ml approximately 12 months after initiation of GFD

   Secondary endpoints
2. Fasting colon volume measured in ml
3. Whole gut transit time measured in hours

Co-variates analysis as indicated above

The basic characteristics of the study population will be calculated using frequencies and proportions.

Objective 1:

For this cohort of patients with newly diagnosed coeliac disease, investigators will compare the mean difference of their fasting small bowel water content (the primary outcome) before and after the initiation of GFD. This will be done using Paired Test at 5% level of significance. This assumes normality of the data, should the data have a high level of skewness non-parametric methods will be used. In order to assess the potential effect modification with age and gender, investigators will stratify the above analysis by those variables. For this purpose age will be considered as categorical variable and analysed as 20 years bands. This analysis will only be conducted for cases with complete follow-up data on MRI scan.

Objectives 2 and 3:

This analysis will be repeated for the two secondary outcomes, namely the volume of the fasting colon and the gastrointestinal transit time.

Co-variate analyses in the coeliac disease group. The potential association between co-variates (gastrointestinal symptoms, Marsh grading etc.) and the three MRI outcomes will be assessed using stepwise linear regression analysis. Investigators will also assess the magnitude of the effect in term of mean difference along with their respective confidence interval. The analysis would be separately conducted for each outcome and co-variates recorded during the first and the subsequent MRI scan.

Should this analysis highlight a few particularly strong associations, investigators will attempt to input those to a regression model to predict either baseline values or change with GFD.

Pilot study in HVs The HVs group is included to provide pilot reference data to inform the design of future studies. Investigators will compare the small bowel water content among the coeliac disease cases to the HVs (controls), and then compare the mean difference pre- and post-measurement between cases and controls using linear regression.

ELIGIBILITY:
Inclusion:

Patients newly diagnosed with coeliac disease:

* Male or female
* Able to give informed consent
* Able to schedule the first MRI scan (Visit 2 of the study) within a month of having had a duodenal biopsy and not yet commenced on a gluten free diet.

Inclusion

Pilot study in healthy volunteers:

* Healthy volunteers (without any comorbidities)
* Able to give informed consent

Exclusion Pilot study in patients

* Any past serious, unstable medical condition, unstable/uncontrolled diabetes mellitus, major psychiatric diagnosis
* Any reported history of gastrointestinal surgery that could affect gastrointestinal function (colectomy, small bowel resection)
* Pregnancy declared by candidate
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Reported alcohol dependence
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test. The following medications can be permitted during the course of the study, as long as they have been used at a constant dosage and were commenced at least 1 month prior to the start of the study: birth control pill, or depot intramuscular contraceptive preparation, oestrogen-progesterone replacement therapy, L-thyroxine, lowdose antidepressants (up to 25 mg day) of amitriptyline, nortriptyline, or selective serotonin reuptake inhibitor), or antihypertensive in the diuretic, angiotensin converting enzyme inhibitor or angiotensin II inhibitor classes. Antibiotic or probiotic treatment in the past 4 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation of any medical trials for the past 3 months
* Judgement by the PI that the candidate who will be unable to comply with the full study protocol e.g. severe COPD
* Noncompliance to gluten free diet after first, untreated MRI.

Exclusion

Healthy volunteers:

Serology positive test for coeliac disease markers

* Any reported history of gastrointestinal surgery that could affect gastrointestinal function (colectomy, small bowel resection)
* Presence of an intestinal stoma
* Pregnancy declared by candidate
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Reported alcohol dependence
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test. The following medications can be permitted during the course of the study, as long as they have been used at a constant dosage and were commenced at least 1 month prior to the start of the study: birth control pill, or depot intramuscular contraceptive preparation, oestrogen-progesterone replacement therapy, L-thyroxine, lowdose antidepressants (up to 25 mg day1 of amitriptyline, nortriptyline, or selective serotonin reuptake inhibitor), or antihypertensive in the diuretic, angiotensin converting enzyme inhibitor or angiotensin II inhibitor classes.
* Proton Pump Inhibitor (PPI), antibiotic or probiotic treatment in the past 12 weeks
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation of any medical trials for the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 36 newly diagnosed coeliac disease patients.
  A parallel group of 36 healthy subjects, frequency matched for age (in 20 years bands) and gender.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Fasting small bowel water content (SBWC) | 12 months
  Fasting small bowel water content (SBWC) measured in ml approximately 12 months after initiation of GFD

SECONDARY OUTCOMES:
Colon volume | 12 months after initiation of gluten free diet
  Fasting colon volume measured in ml
Gut transit time | 12 months after initiation of gluten free diet
  Whole gut transit time measured in hours

OTHER OUTCOMES:
Breath hydrogen | 12 months approximately after recruitment
  Excretion of H2 (hydrogen) gas in breath, measured in parts per million (ppm).

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marciani, PhD, Principal Investigator — University of Nottingham
Locations (1):
- NIHR Biomedical Research Unit in Gastrointestinal and Liver Diseases at Nottingham University Hospitals NHS Trust and the University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Background] Marciani L, Coleman NS, Dunlop SP, Singh G, Marsden CA, Holmes GK, Spiller RC, Gowland PA. Gallbladder contraction, gastric emptying and antral motility: single visit assessment of upper GI function in untreated celiac disease using echo-planar MRI. J Magn Reson Imaging. 2005 Nov;22(5):634-8. doi: 10.1002/jmri.20436. PMID 16193473
- [Background] Hoad CL, Marciani L, Foley S, Totman JJ, Wright J, Bush D, Cox EF, Campbell E, Spiller RC, Gowland PA. Non-invasive quantification of small bowel water content by MRI: a validation study. Phys Med Biol. 2007 Dec 7;52(23):6909-22. doi: 10.1088/0031-9155/52/23/009. Epub 2007 Nov 8. PMID 18029983
- [Background] Pritchard SE, Marciani L, Garsed KC, Hoad CL, Thongborisute W, Roberts E, Gowland PA, Spiller RC. Fasting and postprandial volumes of the undisturbed colon: normal values and changes in diarrhea-predominant irritable bowel syndrome measured using serial MRI. Neurogastroenterol Motil. 2014 Jan;26(1):124-30. doi: 10.1111/nmo.12243. Epub 2013 Oct 17. PMID 24131490
- [Background] Chaddock G, Lam C, Hoad CL, Costigan C, Cox EF, Placidi E, Thexton I, Wright J, Blackshaw PE, Perkins AC, Marciani L, Gowland PA, Spiller RC. Novel MRI tests of orocecal transit time and whole gut transit time: studies in normal subjects. Neurogastroenterol Motil. 2014 Feb;26(2):205-14. doi: 10.1111/nmo.12249. Epub 2013 Oct 25. PMID 24165044
- [Background] Marciani L. Assessment of gastrointestinal motor functions by MRI: a comprehensive review. Neurogastroenterol Motil. 2011 May;23(5):399-407. doi: 10.1111/j.1365-2982.2011.01670.x. Epub 2011 Jan 30. PMID 21276139
- [Derived] Costigan CM, Warren FJ, Duncan AP, Hoad CL, Lewis N, Hill T, Crooks CJ, Morgan PS, Ciacci C, Iovino P, Sanders DS, Hildebrand F, Gowland PA, Spiller RC, Marciani L. One Year of Gluten-Free Diet Impacts Gut Function and Microbiome in Celiac Disease. Clin Gastroenterol Hepatol. 2025 Aug;23(9):1525-1534.e14. doi: 10.1016/j.cgh.2024.11.006. Epub 2024 Dec 9. PMID 39662692
- See also: For more information on the NIHR Biomedical Research Unit in Gastrointestinal and Liver Diseases at Nottingham University Hospitals NHS Trust and the University of Nottingham — http://www.nddcbru.org.uk/